CLINICAL TRIAL: NCT01331395
Title: A Randomized, Controlled Clinical Trial of the Effect of Traditional Chinese Medicine on IVF Success Rates
Brief Title: Effect of Traditional Chinese Medicine on In Vitro Fertilization (IVF) Success Rates
Acronym: TCM-P002
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment rate slower than anticipated.
Sponsor: Pacific Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010.097-1 (Esch)
Record Dates: First submitted 2011-04-04; First posted 2011-04-08 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Primary Female Infertility; Secondary Female Infertility
Keywords: Infertility; IVF; Acupuncture
MeSH Terms: conditions — Infertility | interventions — Medicine, Chinese Traditional; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVF-No Acupuncture (No Intervention): IVF with no Traditional Chinese Medicine: Acupuncture
- IVF-Acupuncture (Active Comparator): IVF with Traditional Chinese Medicine: Acupuncture
  Interventions: Other: Traditional Chinese Medicine

INTERVENTIONS:
Other: Traditional Chinese Medicine — Active arm will receive Acupuncture with their IVF cycle.
  Other Names: Acupuncture
  Arms: IVF-Acupuncture

SUMMARY:
The purpose of this study is to determine the value of combining Traditional Chinese Medicine (TCM) Protocols including acupuncture with In Vitro Fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to understand and provide consent
2. Subject is female, 21-42 years of age at time of screening and has at least one l ovary
3. Subject BMI is > 18 and < 32
4. Subject is experiencing primary or secondary infertility
5. Subject may receive sperm from donated source
6. Subject's partner has sperm in the ejaculate
7. Subject's serum basal FSH is < 11 IU/L
8. Subject's serum basal estradiol level is between 20-80 pg/mL
9. Subject's TSH level is < 3.0 mv/mL
10. Subject's prolactin level is < 24 ng/mL
11. Subject will agree to limit caffeine intake to one cup (76.5 mL/day) by the time of randomization
12. Subject agrees not to make alterations in diet and lifestyle practices other than those that their Medical Practitioner deems necessary in the best interest of the subject
13. Subject agrees not to participate in any other research opportunities for the duration of the study

Exclusion Criteria:

1. Subject is pursuing sex selection
2. Subject is undergoing treatment with an egg donor
3. Subject experienced more than 2 previous failed cycles
4. Subject is undergoing a heparin or lovenox-based protocol
5. Subject is currently taking herbal therapy (1 week wash-out)
6. Subject is currently taking co-interventions of moxibustion and cupping
7. Subject is exhibiting uterine anomalies (i.e.,bicornuate, unicornuate uterus,)
8. Subject is diagnosed with severe endometriosis defined as endometriomas > 4cm
9. Subject is currently receiving acupuncture therapy (Subject must agree to a 30 day washout period prior to randomization)
10. Subject has history of recurrent spontaneous abortions defined as > 3
11. Subjects with a Beck Depression Inventory (BDI-II) of 29 or higher at screening, indicative of severe depression, will be excluded from the study and referred for further psychological evaluation by our in-house licensed mental health professional.

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who receive an embryo transfer which results in a live birth. | Average of 1 year
  Embryo transfer resulting in Live Birth up to 40 weeks gestation
The proportion of subjects in the active treatment group experiencing no SAE's attributable to ACU. | Overall to be collected at interim analysis of 138 subjects and at study completion of 276 patients

SECONDARY OUTCOMES:
1. The proportion of subjects who undergo an embryo transfer which results in implantation as evidenced by USS at 7 weeks. | Average of 4 months
  At 7 week ultrasound
Effect of the IVF/ICSI treatment on quality of life and psychological factors assessed with the Fertility Quality of Life Questionnaire (FertiQoL 2008) and the Spielberger State Trait Anxiety Inventory (STAI). | Average of two months
  Repeat measures at Screening, Treatment Month and at Embryo Transfer

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Schriock, MD, Principal Investigator — Pacific Fertility Center

REFERENCES:
- See also: Related Info — http://www.pacificfertilitycenter.com/